CLINICAL TRIAL: NCT06003595
Title: Long-term Outcome After Removal of Rib Stabilization Hardware in Patients With Blunt Chest Trauma
Acronym: REMOVE
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-01191; kt23Lardinois3
Record Dates: First submitted 2023-07-18; First posted 2023-08-22 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Rib Fractures
Keywords: surgical stabilization of rib fractures (SSRF); hardware failure; hardware-related complications; hardware removal; blunt chest trauma; rib osteosynthesis
MeSH Terms: conditions — Rib Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Surgical stabilization of rib fractures (SSRF) and subsequent hardware removal: Patients treated at the Department of Thoracic Surgery at the University Hospital Basel between 01.09.2017 and start date Remove Study with a diagnosis of rib fracture and with surgical stabilization of rib fracture and subsequent hardware removal will be identified.
  Interventions: Other: Data collection on patient reported long-term outcome of SSRF hardware removal

INTERVENTIONS:
Other: Data collection on patient reported long-term outcome of SSRF hardware removal — One prospective follow-up visit will be performed. On this visit the patient reported long-term outcome will be documented through a health survey.

SUMMARY:
The main study objective is to evaluate the long-term outcome in a prospective follow-up visit of patients who underwent hardware removal after surgical stabilization of rib fractures (SSRF) after a blunt chest trauma .

DETAILED DESCRIPTION:
Potential of surgical stabilization of rib fractures (SSRF) to improve clinical outcomes in patients has been demonstrated with increasing interest of surgeons in this procedure and indications for SSRF expanding. Some reports found signals for hardware removal after SSRF such as hardware failure, infections and persisting pain. There is currently lack of studies collecting systematically long-term outcomes after SSRF hardware removal. For that reason, this project presents the retrospective case series of patients with removal of osteosynthetic material after rib stabilisation treated at Department of Thoracic Surgery of the University Hospital Basel (USB). The recovery of these patients will be reviewed and a prospective evaluation of long-term outcomes will be done. The aim is to provide an insight and implications for treatment strategies of future patients. Most of the collected patient data are retrospective data. One prospective follow-up visit inclusive a health survey per patient will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Patient treated at the Department of Thoracic Surgery, USB for implantation and removal of rib fixation hardware
* Blunt chest trauma/injuries to the thorax: Patient with blunt chest trauma (with or without polytrauma) before SSRF implantation and subsequent hardware removal
* Rib fracture: At least one rib fracture (unilateral and/or bilateral incl. flail chest) on radiography chest imaging on time of SSRF implantation. Patients with rib fracture/non-union due to pseudoarthrosis are included.
* Rib fixation material implantation and removal: Patient underwent surgery for rib fracture and implantation of at least one (partially or complete) rib fixation material (at any time point) with later hardware removal (partially or complete) (at any time point between 01.09.2017 and 30.09.2023)
* Patient of all gender
* Patient ≥18 years at time point of rib stabilization
* Signed written informed consent prior to initiation of any protocol-specific activities/procedure
* Patient will be included if a signed USB general research consent approval is available but patient cannot be reached or disagreed to come to the follow-up visit
* Patient who died will be included if a signed USB general research consent approval is available

Exclusion Criteria:

* Patients who received re-osteosynthesis on the same day as hardware removal
* Patients received conservative therapy or surgery with absorbable plates
* On hardware implantation:

  * Penetrating chest trauma
  * Only random findings of rib fractures
  * Solitary sternocostal joint fracture and/or solitary sternum fracture and/or solitary fractures of rib connecting parts and/or solitary thoracic spine/vertebra fracture
  * In-hospital: Patient suffered only iatrogenic rib facture during a surgery, cardiac surgery
  * Rib fractures/non-unions caused by malignancy or rib surgery due to malignancy, radiation therapy, COPD, coughing
* Inability to follow procedures or insufficient knowledge of language (German/French) or impaired communication or inability to give consent
* Patients who have clearly stated that they would not agree in providing their clinical data for scientific purposes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with blunt chest trauma who underwent hardware removal after rib stabilisation between September 01, 2017 and September 30, 2023. The patients received hardware implantation and hardware removal at the Department of Thoracic Surgery of the University Hospital Basel.
Sampling Method: Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2023-08-04 (Actual); Primary Completion 2024-01-08 (Actual); Study Completion 2024-01-08 (Actual)

PRIMARY OUTCOMES:
Health survey of long-term outcome after hardware removal (Quality of life assessment) | One time assessment at baseline (prospective Follow up-visit)
  The questions are formulated as an adapted question set of the EQ-5D-5L Dimension (EQ-5D-5L) questionnaire followed by additional study specific questions. A numerical rating scale (NRS) will be used for evaluation from 0 - 10. In addition, the patient will be asked to rate the condition now compared to before hardware removal in four categories (less good, no change, slightly better, much better). The analysis of the project data will be done descriptive.

SECONDARY OUTCOMES:
Number of removed hardware | Up to 3 years until prospective Follow up-visit
  Number of removed hardware and affected ribs (retrospective analyses)
Number of broken and fixed ribs | Up to 3 years until prospective Follow up-visit
  Number of broken and fixed ribs with used hardware (retrospective analyses)
Interval between SSRF and hardware removal | Up to 3 years until prospective Follow up-visit
  Interval between SSRF and hardware removal (retrospective analyses)
Interval between SSRF and follow-up visit | Up to 3 years until prospective Follow up-visit
  Interval between SSRF and follow-up visit (retrospective analyses)
Occurrence of significant complications during and 30 days after SSRF hardware removal | Up to 3 years until prospective Follow up-visit
  Occurrence of significant complications during and 30 days after SSRF hardware removal (retrospective analyses)
Surgical indication for hardware removal | Up to 3 years until prospective Follow up-visit
  Surgical indication for hardware removal

CONTACTS AND LOCATIONS:
Overall Officials: Maria Stepankova, MD, Principal Investigator — Department of Thoracic Surgery, University Hospital Basel
Locations (1):
- Department of Thoracic Surgery, University Hospital Basel, Basel, Switzerland

REFERENCES:
- [Result] Svec MB, Bachmann H, Hojski A, Macharia-Nimietz EF, Dackam SVC, Lardinois D. Long-term outcomes after removal of rib stabilization hardware in patients with blunt chest trauma. Eur J Trauma Emerg Surg. 2025 Apr 29;51(1):187. doi: 10.1007/s00068-025-02858-y. PMID 40299046